CLINICAL TRIAL: NCT04145934
Title: A Randomized Controlled Trial of a Multicomponent Walking Aid Program for People With MS
Acronym: ADSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Cameron, Neurologist, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20191
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: fall prevention; walking aid; physical therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training (Experimental): The subjects receive the ADSTEP intervention
  Interventions: Behavioral: ADSTEP
- waitlist (No Intervention): These subjects receive two brochures on fall prevention and walking aid selection, and a letter is sent to their care provider informing them that the subject has reported falling. Subjects in this group will be offered the ADSTEP intervention once their study participation is complete.

INTERVENTIONS:
Behavioral: ADSTEP — ADSTEP is a training program of six weekly one-on-one sessions with a physical therapist intended to reduce falls among people who use a hand-held walking aid, such as a cane or a walker. ADSTEP focuses on training in the use of the walking aid, and includes gait evaluation, walking aid selection and fitting, and progressive task-oriented training with the walking aid.
  Arms: training

SUMMARY:
This is a randomized controlled trial of the Assistive Device Selection, Training, and Education Program (ADSTEP). ADSTEP is a training program of six weekly one-on-one sessions with a physical therapist intended to reduce falls among people who use a hand-held walking aid, such as a cane or a walker. ADSTEP focuses on training in the use of the walking aid, and includes gait evaluation, walking aid selection and fitting, and progressive task-oriented training with the walking aid.

Participants will be randomized to receive ADSTEP or a waitlist control intervention; those in the control condition will receive National MS Society brochures on fall prevention and walking aid selection, and a letter will be sent informing their care provider that the subject reports falling. All subjects will complete an assessment visit at baseline, and follow-up assessments at about 8 weeks and about 6 months after that. Subjects will complete paper questionnaires of patient reported outcomes (PROs), a modified Functional Gait Assessment / Dynamic Gait Index, and will track fall sustained over their participation in the study using monthly paper fall calendars. At the end of study participation, all subjects in the control group will be offered the opportunity to receive ADSTEP.

ELIGIBILITY:
Inclusion Criteria:

1. A definite diagnosis of MS of any type;
2. 18 years of age or older;
3. Self-reported history of at least one fall in the previous year;
4. Ability to walk at least 25 feet with or without an assistive device;
5. Intermittent or constant unilateral or bilateral assistance required to walk;
6. No MS exacerbations for the past 30 days;
7. Willingness to complete a written daily record of falls for about 8 months.

Exclusion Criteria:

1. Currently receiving physical therapy, or having any plans to receive physical therapy in the upcoming 8 months (duration of study participation);
2. Serious psychiatric or medical conditions that would preclude reliable participation in the study (e.g. dementia, deafness, blindness);
3. Inability to follow directions in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Reported Falls at 8 months | daily for 8 months
  Paper Fall Calendars

SECONDARY OUTCOMES:
Change from Baseline in Functional Gait Assessment / Dynamic Gait Index | At baseline, 8 weeks, and 8 months
  Functional Gait Assessment / Dynamic Gait Index

OTHER OUTCOMES:
Change from Baseline in Walking Aid Satisfaction | At baseline, 8 weeks, and 8 months
  Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0)
Change from Baseline in Physical Activity | At baseline, 8 weeks, and 8 months
  International Physical Activity Questionnaire (IPAQ)
Change from Baseline in Walking Ability | At baseline, 8 weeks, and 8 months
  Multiple Sclerosis Walking Scale-12 (MSWS-12). Min/max score: 12/60, higher indicates worse outcome
Change from Baseline in Quality of Life | At baseline, 8 weeks, and 8 months
  Multiple Sclerosis Impact Scale-29 (MSIS-29). Min/max score: 29/145, higher indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cameron, PT, MD, MCR, Principal Investigator — Oregon Health & Science University / VA Portland Health Care System
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All data obtained will be placed in a data repository maintained at the VA Portland Health Care System. Data in the repository will be accessible to other researchers at the discretion of the repository director, upon execution of a data use agreement.
Time Frame: Data will become available shortly after completion of data collection (anticipated for December 2021). Data will be available indefinitely thereafter.
Access Criteria: Execution of a data use agreement with VA Portland Health Care System